CLINICAL TRIAL: NCT02497625
Title: Effectiveness of the Addition of Therapeutic Alliance to Minimal Intervention Treatment for Chronic Low Back Pain With Low Risk of Psychosocial Factors: a Randomized Controlled Trial
Brief Title: Effectiveness of Therapeutic Alliance and Minimal Intervention for Chronic Low Back Pain
Acronym: TalkBack
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Cidade de Sao Paulo (Other)
Responsible Party: Principal Investigator, Cristina Maria Nunes Cabral, Professor PhD, Universidade Cidade de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 44720315.5.0000.5372
Record Dates: First submitted 2015-07-10; First posted 2015-07-14 (Estimated); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Low Back Pain
Keywords: Low back pain; Empathy; Subgroups; Minimal intervention
MeSH Terms: conditions — Low Back Pain | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Positive Therapeutic Alliance (Experimental): Intervention involving reassurance and information related to the return to daily activities, advice on dealing with the pain and clear explanation of signs and symptoms. The session will take 60 minutes and will be structured to increase the therapeutic alliance and empathy. Patients will be instructed to return in a week for further consultation to clarify doubts.
  Interventions: Behavioral: Positive Therapeutic Alliance
- Usual Care (Active Comparator): Information about low back pain based on Back Book. The therapy will be performed with limited interaction between patient and therapist and the information will be transmitted in a clear and direct way. The limited interaction between patient and therapist in this group will be established at the first session lasting 45-60 minutes. Patients will be instructed to return for a visit after a week to clarify questions.
  Interventions: Behavioral: Usual care
- Control group (Other): Patients will not receive intervention in the first mo nth of enrollment. After a year, the treatment offered to the Positive Therapeutic Alliance or Usual Care group will be available for patients who are interested.
  Interventions: Other: Control group

INTERVENTIONS:
Behavioral: Positive Therapeutic Alliance — Intervention involving reassurance and information related to the return to daily activities, advice on dealing with the pain and clear explanation of signs and symptoms. The session will take 60 minutes and will be structured to increase the therapeutic alliance and empathy. Patients will be instructed to return in a week for further consultation to clarify doubts.
  Arms: Positive Therapeutic Alliance
Behavioral: Usual care — Information about low back pain based on Back Book. The therapy will be performed with limited interaction between patient and therapist and the information will be transmitted in a clear and direct way. The limited interaction between patient and therapist in this group will be established at the first session lasting 45-60 minutes. Patients will be instructed to return for a visit after a week to clarify questions.
  Arms: Usual Care
Other: Control group — Patients will not receive intervention in the first month in which they are enrolled. After a year, the treatment offered to the Positive Therapeutic Alliance or Usual Care group will be available for patients who are interested.
  Arms: Control group

SUMMARY:
This study aims to evaluate the effectiveness of minimal intervention and therapeutic alliance in pain, specific and general disability, global perceived effect, empathy, credibility and expectation of improvement in patients with chronic non-specific low back pain

DETAILED DESCRIPTION:
Low back pain remains a global public health problem. The classification of patients in low back pain subgroups aims to optimize the health system and provide the quantity and the type of proper technique for each patient. Several factors may influence physical therapy. The therapeutic alliance may be defined as harmony or social connection between the therapist and the patient and may influence the treatment effect. The aim of this study is to evaluate the effectiveness of the addition of the therapeutic alliance to a minimum intervention for the treatment of chronic non-specific low back pain with low risk of psychosocial factors.

ELIGIBILITY:
Inclusion Criteria

* Patients waiting for treatment in the waiting list of physical therapy clinics
* Diagnosis of chronic non-specific low back pain (over 12 weeks)
* More than 18 years
* Able to read and write the Portuguese language
* Low risk of psychosocial factors (less than 3 points in the STarT Back Screening Tool).

Exclusion criteria

* Spine surgery history
* Nerve root compromise
* Cognitive impairment related disorders
* Pregnants

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2015-09; Primary Completion 2017-06-30 (Actual); Study Completion 2021-02-11 (Actual)

PRIMARY OUTCOMES:
Pain intensity | One month after randomization
  Pain intensity will be measured by an 11-point Pain Numerical Rating Scale
Specific disability | One month after randomization
  Specific disability associated with low back pain will be measured by the 11-point Patient Specific Functional Scale.

SECONDARY OUTCOMES:
Pain intensity | Six and twelve months after randomization
  Pain intensity will be measured by an 11-point Pain Numerical Rating Scale
Specific disability | Six and twelve months after randomization
  Specific disability associated with low back pain will be measured by the 11-point Patient Specific Functional Scale.
Disability | One, six and twelve months after randomization
  Disability associated with low back pain will be measured by the 0-100 scale of the Oswestry Disability Index
Global impression of recovery | One, six and twelve months after randomization
  Global impression of recovery will be measured by an 11-point Global Perceived Effect Scale

OTHER OUTCOMES:
Empathy | One week after the first session of treatment
  Empathy will be measured by a 50-point scale of the Consultation and Relational Empathy (CARE) questionnaire
Credibility | After the first session of treatment
  The credibility regarding the treatment will be evaluated using 0-24 point scale.
Expectation of improvement | One week after the first session of treatment
  The expectation of improvement will be assessed with a numerical scale of 11 points

CONTACTS AND LOCATIONS:
Overall Officials: Felipe RC Fagundes, MsC, Principal Investigator — Universidade Cidade de São Paulo
Locations (1):
- Physical Therapy Outpatient Department, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fagundes FR, de Melo do Espirito Santo C, de Luna Teixeira FM, Tonini TV, Cabral CM. Effectiveness of the addition of therapeutic alliance with minimal intervention in the treatment of patients with chronic, nonspecific low back pain and low risk of involvement of psychosocial factors: a study protocol for a randomized controlled trial (TalkBack trial). Trials. 2017 Jan 31;18(1):49. doi: 10.1186/s13063-017-1784-z. PMID 28143504